CLINICAL TRIAL: NCT00487331
Title: Acupuncture for Treatment of Uncontrolled Pain: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-1113
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2013-10

CONDITIONS: Solid Tumors; Pain
Keywords: Solid Tumors; Acupuncture; Uncontrolled Pain; Pain
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): Acupuncture sessions 1-3 times per week. 2 pain questionnaires + satisfaction survey completed at beginning and end of treatment.
  Interventions: Other: Acupuncture; Behavioral: Survey

INTERVENTIONS:
Other: Acupuncture — Acupuncture sessions 1-3 times per week.
Behavioral: Survey — 2 pain questionnaires + satisfaction survey completed at beginning and end of treatment
  Other Names: questionnaire

SUMMARY:
The goal of this clinical research study is to learn if using acupuncture with or without electrical stimulation in cancer patients with high levels of pain can help to relieve the pain.

DETAILED DESCRIPTION:
Acupuncture involves the insertion of small, solid, sterile needles into specific points on the skin. The needles are placed in areas that are intended to help relieve pain. Electrical stimulation is often applied to the needles to improve the treatment effects. The procedure is designed to be comfortable and relaxing.

Acupuncture Sessions:

If you are found to be eligible to take part in this study, you will receive acupuncture sessions 1-3 times per week in the acupuncture clinic at M. D. Anderson. The number of sessions will depend on the type and location of the pain you may be experiencing.

For each session, you will be placed in a comfortable position and the study doctor/acupuncturist will find points on your body and/or ears where the needles will be placed. These points will be chosen based on the symptoms you are having at the time of treatment, the location of the pain, and the type of pain.

Very thin, solid, sterile, stainless steel needles will be used. All of the needles are specially made for acupuncture. The depth of the needle in the skin, the number of needles, and whether the needles are near or far from the areas of pain will vary from person to person, based on standard acupuncture procedures.

In most instances, needles placed on body points will remain in place for about 20-30 minutes. This length of time is the same for some points on the ears as well, but in some instances, small gold or stainless steel needles may be placed on the ears. These needles for the ears are designed to remain in place for 3-4 days. The ear needles are slightly larger than the head of a pin and have a small ridge that is designed to help them remain in place. If you prefer, a small flesh colored adhesive patch can be placed over the ear needles as added protection. This is usually not necessary, but can be added if you prefer.

Electrical stimulation may be added to some of the needles, depending on the type of pain you are experiencing and where it is located. This involves placing wires on the needles, which are connected to a machine that delivers a mild electrical current through the wires. The intensity (strength) of the electrical current will be adjusted gradually until it is at a comfortable level for you.

Study Procedures:

At each session, before you receive the acupuncture, the following procedures will be performed:

* Your vital signs will be measured.
* You will be asked about any medications you may be taking and any side effects you may be experiencing.
* The color and coating of your tongue and the quality of your pulse will be recorded.
* If you are receiving medications that are known to affect your blood counts, blood (about 1 teaspoon) will be drawn for routine tests to check your blood counts.

Each study visit will last about 1 hour. During the study, you may still receive your regular pain treatments outside of this study.

Length of Study Participation:

You may receive up to 10 acupuncture sessions (depending on the location and type of pain). If intolerable side effects or symptoms occur, you will be taken off study early.

End-of-Study Visit:

On the day of your last acupuncture session (called the end-of-study visit), or if you go off study early for any reason, the following procedures will be performed:

Your medical history will be recorded. Your vital signs will be measured. You will be asked about any medications you may be taking and any side effects you may have experienced.

You will complete the same 2 pain questionnaires as before. You will also complete a questionnaire that has questions about your level of satisfaction with the acupuncture services that were provided. In total, the 3 questionnaires should take about 15 minutes to complete.

Your tongue and pulse will be evaluated.

Study Completion:

After the end-of-study visit, your participation in this study will be over.

This is an investigational study. The needles used in this study are FDA approved for use in patients with cancer. It is considered experimental, however, to provide acupuncture services to patients with cancer who have uncontrolled pain. Up to 64 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, or the legal guardians of patients must have the ability to understand English, sign a written informed consent, and be willing to follow protocol requirements.
2. ECOG Performance Status of 0, 1, or 2.
3. Pain score >/= 4 on the on a 0-10 NRS pain scale after all efforts have been attempted in the PMC to control pain.

Exclusion Criteria:

1. Local infection at or near the acupuncture site. (Although acupuncture is a minimally invasive procedure, patients will be excluded if there is an indication of infection.)
2. Deformities that could interfere with accurate acupuncture point location.
3. Known coagulopathy and taking any dose of warfarin (i.e., Coumadin) or heparin, including low molecular weight heparin (i.e., Lovenox). Patients may participate if they are taking Plavix, aspirin or other non-steroidal anti-inflammatory agents.
4. Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry as these patients may not be able to cooperative with this slightly invasive procedure or with the data collection process.
5. Labs: platelets <100,000 and/or WBC < 3000 on most recent report. (Note: Whether or not lab work is drawn prior to beginning the acupuncture treatment will be left to the discretion of the referring physician. Patients with platelets <100,000 may participate with written approval from the attending physician.)
6. Planned changes in the pain medication regimen.
7. Women who are pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Patients' Reported Satisfaction with Acupuncture Services | Derived from surveys completed by participating patients over 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Larry C. Driver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org